CLINICAL TRIAL: NCT06074666
Title: Behavioral Parenting Skills as a Novel Target for Improving Pediatric Medication Adherence: Study 3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I 3774823; R01CA258337 (NIH)
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Acute Lymphoblastic Leukemia, Pediatric
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CareMeds Intervention (Experimental): Participants complete the CareMeds parent training sessions during weeks 2, 3 and 4.
  Interventions: Behavioral: CareMeds Intervention
- Usual Care (Active Comparator): Usual care consists of medical consultations and supportive care, The usual care group will serve as a delayed intervention/wait list group for which 3 parent training sessions will be offered during weeks 13 through 15.
  Interventions: Behavioral: Usual Care Group

INTERVENTIONS:
Behavioral: CareMeds Intervention — 3 parenting sessions will be offered during weeks 2 through 4 of the study period.
  Arms: CareMeds Intervention
Behavioral: Usual Care Group — 3 parenting sessions will be offered during weeks 13 through 15 of the study period.
  Arms: Usual Care

SUMMARY:
The current study will assess the acceptability and feasibility of the CareMeds intervention with a larger sample (N = 100) across multiple sites in Buffalo, NY, and Atlanta, GA.

DETAILED DESCRIPTION:
This is a pilot randomized controlled trial of the CareMeds program to assess feasibility and obtain preliminary efficacy data among families of young children (ages 3-9) with ALL. The objective of this aim is to implement our study procedures and study conditions (CareMeds vs. usual care control). We hypothesize that pilot findings will support the feasibility of the intervention and suggest important improvements in our behavioral secondary outcomes (i.e., behavioral parenting skills, medication adherence

ELIGIBILITY:
Inclusion Criteria:

* Parent of a child who is diagnosed and being treated for any type of acute lymphoblastic leukemia (ALL) at a study site.
* Parent has primary medication responsibility.
* Pediatric patient aged 3-9 years
* Child on therapy that includes home-based oral anti-cancer medication taken at home, such as 6-MP.
* Parent has verbal English or Spanish fluency.
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Parent of a child who is not diagnosed nor being treated for any type of acute lymphoblastic leukemia (ALL) at a study site.
* Parent does not have primary medication responsibility.
* Pediatric patient aged 3-9 years
* Pediatric patient is not on therapy that includes oral anti-cancer medication (e.g., 6-MP).
* Parent does not have verbal English or Spanish fluency.
* Parent is unwilling or unable to follow protocol requirements

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the CareMeds 3 sessions | up to 3 years
  enrollment rates will be measured by number of consents . Reasons for refusal will also be captured

SECONDARY OUTCOMES:
Behavioral Parenting skills | Weeks 1, 4 and 12.
  Self reported measure to assess the frequency of parental engagement on a scale from 1 (not at all) to 7 (Most of the time)
Oral Chemotherapy adherence | UP to week 12
  Will be measured by the number of days with MEMS cap openings to the number of days 6-MP was prescribed.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Bouchard, PhD, Principal Investigator — Roswell Park Comprehensive Cancer Center
Locations (1):
- Roswell Park Comprehensive Cancer Center, Buffalo, New York, United States